CLINICAL TRIAL: NCT01053507
Title: Evaluation of the Efficacy of Treximet for Prevention of Post Traumatic Headache Associated With Cognitive Dysfunction
Brief Title: Treximet for Prevention of Post Traumatic Headache Associated With Cognitive Dysfunction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment rate was slower than anticipated.
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 114126
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Post-Traumatic Headache
Keywords: Headache; Post-traumatic headache; Brain injury; Cognitive impairment
MeSH Terms: conditions — Post-Traumatic Headache; Headache; Brain Injuries; Cognitive Dysfunction | interventions — Sumatriptan; Naproxen; sumatriptan-naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treximet (Active Comparator): In the 30-day Treatment Period, subjects randomized to Treximet will treat with 1 tablet Treximet (sumatriptan 85mg / naproxen sodium 500mg) per day x 30 days.
  Interventions: Drug: sumatriptan/naproxen sodium
- Placebo (Placebo Comparator): In the 30-day Treatment Period, subjects randomized to placebo will treat with 1 tablet placebo x 30 days. Placebo matches Treximet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: sumatriptan/naproxen sodium — Each tablet of Treximet for oral administration contains sumatriptan 85mg / naproxen sodium 500mg. Study medication is to be administered 1 tablet per day at the same time each day x 30 days in the Treatment Period.
  Other Names: Treximet
  Arms: Treximet
Drug: Placebo — Each tablet of placebo for oral administration matches Treximet. Placebo is to be administered 1 tablet per day at the same time each day x 30 days in the Treatment Period.
  Arms: Placebo

SUMMARY:
This study will evaluate the effectiveness of Treximet when taken for post traumatic headache by measuring any change in the number of headache days or any change in a subject's ability to think following treatment with study medication. Eligible subjects will complete 3 visits. Following Visit 1, subjects will treat with their usual medication and document headache symptoms and therapy in a Headache Diary. After 30 days, subjects will return for Visit 2 and be randomized (like the flip of a coin) to receive Treximet or matching placebo to treat at the same time each day. Treximet will be provided to treat any headache that occurs. Subjects will complete a daily Diary. After 30 days, subjects will exit the study at Visit 3.

DETAILED DESCRIPTION:
Subjects will be enrolled at 3 investigative sites. At Visit 1, a medical, headache, and medication history will be collected and a physical and neurological exam with vital signs will be performed. An ECG will be completed if one has not been completed in the previous 6 months. Subjects will be administered a series of psychological tests to help the study doctor decide whether or not a subject is eligible. The Headache Impact Test-6 and Migraine Specific Quality of Life Questionnaire will be completed at each visit. During a 30-day Baseline Period, subjects will treat with their usual medication and complete a daily Diary documenting headache symptoms and treatment. At Visits 2 and 3 subjects will complete the Mental Efficiency Workload Test and Migraine Early Warning Tool. Following randomization at Visit 2, subjects will treat daily for 30 days with Treximet or a matching placebo. Subjects will be provided with Treximet for rescue of any persisting or recurring headache. During the Treatment Period, subjects will complete a daily Diary reporting headache symptoms and response to treatment. After the 30-day Treatment Period, subjects will exit the study at Visit 3 .

ELIGIBILITY:
Inclusion Criteria:

Subject

* is male or female between the ages of 18-65. A female is eligible to enter and participate in this study if she is of: a.non-childbearing potential (i.e., physiologically incapable of becoming pregnant); or,b. child-bearing potential, has a negative pregnancy test (urine or serum) at Visit 2, and agrees to one of the following: Complete abstinence from intercourse from 2 weeks prior to administration of the investigational product, throughout the study, and for a time interval (5 days) after completion or premature discontinuation from the study to account for elimination of the investigational drug; subjects utilizing this method must agree to use an alternate method of contraception if they should become sexually active and will be queried on whether they have been abstinent when they present to the clinic for the final visit or, Female sterilization; or, Sterilization of male partner; or, Implants of levonorgestrel; or, Injectable progestogen; or, Oral contraceptive (combined or progestogen only); or, Any intrauterine device (IUD) with published data showing that the highest expected failure rate is less than 1% per year (not all IUDs meet this criterion); or, Spermicide plus a mechanical barrier (e.g., spermicide plus a male condom or a female diaphragm); or, Any other barrier methods (only if used in combination with any of the above acceptable methods); or, Any other methods with published data showing that the highest expected failure rate for that method is less than 1% per year.
* is formally diagnosed with International Classification of Headache Disorders (ICHD) 5.2.2 chronic post traumatic headache
* has >15 headache days per month in past 3 months
* has headache that, if left untreated, would have at least 1 symptom of migraine (nausea, vomiting, photophobia, or phonophobia) or respond to a triptan or ergotamine-containing medication with at least 50% of headaches
* is medically stable as determined by the Investigator
* if taking a headache preventive medication, has been on a stabilized dosage for at least 30 days prior to screening.
* if taking any concomitant medications, is on a stabilized dosage at the discretion of the investigator
* has chronic headache history only after the traumatic brain injury (TBI)
* is able to understand and communicate intelligibly with the study observer
* is able to take oral medication, adhere to the medication regimens and perform study procedures
* is able to read and comprehend written instructions and be willing to complete all procedures and assessments required by this protocol
* is able to demonstrate the willingness to participate by signing and understanding an informed consent after full explanation of the study
* has self-reported cognitive inefficiency or "brain-fog" during headache

Exclusion Criteria:

Subject

* has a history of serotonin syndrome
* has any medical condition that, in the opinion of the investigator, could alter the response to study medication or confound the results of the study
* is female of childbearing potential not using adequate contraceptive measures
* has history of retinal, basilar or hemiplegic migraine, cluster headache, or secondary headaches (such as due to infection, alterations of homeostasis, ear nose and throat (ENT) or psychiatric disorders, cranial or cervical disorders or neuralgias)
* in the investigator's opinion, is likely to have unrecognized cardiovascular or cerebrovascular disease (based on history or the presence of risk factors including but not limited to, hypertension, hypercholesterolemia, smoker, obesity, diabetes, or family history of coronary artery disease)
* has blood pressure ≥140/90 millimeters of mercury (mmHg) in 2 out of 3 BP measurements at screening or is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker
* has a history of significant congenital heart disease, cardiac arrhythmias requiring medication, or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study
* has evidence or history of any ischemic vascular diseases including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome, or signs/symptoms consistent with any of the above
* has evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower the convulsive threshold; or has been treated with an antiepileptic drug for seizure control within 5 years prior to screening
* has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study
* has hypersensitivity, intolerance, or contraindication to the use of any triptan, nonsteroidal antiinflammatory drug (NSAID) or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma
* is currently taking, or has taken in the previous three months, a migraine prophylactic medication containing methysergide; or is taking a migraine or menstrual migraine prophylactic medication that is not stabilized (i.e. start or change of dose within 30 days prior to screening)
* has a recent history of regular use of opioids or barbiturates for treatment of their migraine headache and/or other non-migraine pain or any medication overuse that in the opinion of the investigator has exacerbated or contributed to the current headache pattern of the subject.
* has taken, or plans to take, a monoamine oxidase inhibitor (MAOI), including herbal preparations containing St. John's Wort (Hypericum perforatum), anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
* has history of any bleeding disorder or is currently taking any anti-coagulant or any antiplatelet agent.
* has evidence or history of any gastrointestinal surgery or GI ulceration or perforation in the past six months, gastrointestinal bleeding in the past year; or evidence or history of inflammatory bowel disease
* is pregnant, actively trying to become pregnant, or breast feeding
* has evidence of alcohol or substance abuse within the last year or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial.
* has participated in an investigational drug trial within the previous four weeks or plans to participate in another study at any time during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (3):
- United States (3):
  - Clinvest, Springfield, Missouri
  - Nashville Neuroscience Group, PC, Nashville, Tennessee
  - Scott & White Memorial Hospital and Clinic, Temple, Texas

REFERENCES:
- [Background] Baandrup L, Jensen R. Chronic post-traumatic headache--a clinical analysis in relation to the International Headache Classification 2nd Edition. Cephalalgia. 2005 Feb;25(2):132-8. doi: 10.1111/j.1468-2982.2004.00818.x. PMID 15658950
- [Background] Headache Classification Subcommittee of the International Headache Society. The International Classification of Headache Disorders: 2nd edition. Cephalalgia. 2004;24 Suppl 1:9-160. doi: 10.1111/j.1468-2982.2003.00824.x. No abstract available. PMID 14979299
- [Background] Cady R, Farmer K. Soft tissue injuries: diagnosis and treatment. Posttraumatic headache. In Windsor R, Lox D (eds.) Hanley and Belfus, Inc. Philadelphia, PA. 207-224.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treximet | Placebo
Started | 11 | 12
Completed | 8 | 11
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treximet | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.36 (9.83) | 35.83 (12.01) | 38.48 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Headache Days
Description: Change in number of headache days at Day 0 vs. Day 30 in Treximet arm vs. Placebo arm.
Time Frame: Day 0, Day 30
Population: Analysis population only includes subjects that provided data at both time points (Day 0 and Day 30).
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treximet | Placebo
Number analyzed (Participants) | 7 | 10
days | -3.00 (7.6) | -0.30 (5.3)

2. Primary Outcome: Change in Number of Associated Headache Symptoms
Description: Change in number of associated headache symptoms at Day 0 vs. Day 30 in Treximet arm vs. Placebo arm. Associated headache symptoms measured included number of incidences of: sleeplessness, difficulty thinking, and bodily pain.
Time Frame: Day 0, Day 30
Population: Analysis population only includes subjects that provided data at both time points (Day 0 and Day 30).
Measure: Mean (Standard Deviation); unit: change in number of symptoms
Arm/Group | Treximet | Placebo
Number analyzed (Participants) | 7 | 10
change in number of symptoms
  Change in Sleeplessness | 2.43 (7.76) | -2.30 (3.47)
  Change in Difficulty Thinking | 0.14 (12.32) | 0.00 (4.83)
  Change in Bodily Pain | -1.71 (6.52) | -3.80 (5.67)

3. Secondary Outcome: Mental Efficiency Workload Test (MEWT) Performance Index
Description: The Mental Efficiency Workload Test (MEWT) performance index is a scale with minimum and maximum values of 1 to 10, 1 indicates the poorest level and 10 indicates the best level of cognitive functioning.
Time Frame: Day 0, Day 30
Population: Analysis population only includes subjects that provided data at both time points (Day 0 and Day 30).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treximet | Placebo
Number analyzed (Participants) | 6 | 9
units on a scale
  Day 0 | 3.10 (2.28) | 3.4 (2.27)
  Day 30 | 3.17 (2.23) | 3.11 (2.09)

4. Secondary Outcome: Headache Impact Test-6 (HIT-6) Score
Description: The Headache Impact Test-6 (HIT-6) scale measures the impact of headache symptoms on subject's life. Possible scores range from 36 to 78. Score of 48 or less indicates headache has little impact on life. Score of 60-78 indicative of very severe impact.
Time Frame: Day 0, Day 30
Population: Analysis population only includes subjects that provided data at both time points (Day 0 and Day 30).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treximet | Placebo
Number analyzed (Participants) | 7 | 11
units on a scale
  Day 0 | 59.43 (6.65) | 61.91 (3.21)
  Day 30 | 58.57 (6.13) | 61.91 (6.44)

5. Secondary Outcome: Migraine Specific Quality of Life Questionnaire (MSQ)
Description: The Migraine-Specific Quality of Life Questionnaire (MSQ) is a scale that measures the impact of migraine across three aspects: role function-restrictive (RR), role function-preventive (RP), and emotional function (EF). Possible scores on each subscale range from a 0 to 100 scale such that higher scores indicate better quality of life.
Time Frame: Day 0, Day 30
Population: Analysis population only includes subjects that provided data at both time points (Day 0 and Day 30).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treximet | Placebo
Number analyzed (Participants) | 7 | 11
units on a scale
  Day 0 - Role Function-Restrictive Score | 60 (12.34) | 45.71 (16.95)
  Day 30 - Role Function-Restrictive Score | 59.59 (23.81) | 50.39 (19.35)
  Day 0 - Role Function-Preventive Score | 79.29 (14.84) | 68.64 (22.81)
  Day 30 - Role Function-Preventive Score | 80 (13.84) | 69.55 (24.95)
  Day 0 - Emotional Function Score | 60 (18.05) | 50.91 (25.69)
  Day 30 - Emotional Function Score | 65.03 (28.76) | 57.58 (29.25)

ADVERSE EVENTS:
Time Frame: Day 0, Day +30
Arm/Group | Treximet | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 7/11 | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treximet (N=11) | Placebo (N=12)
Throat Tightness (Gastrointestinal disorders) | 0 (0) | 1 (8)
Chest Pressure (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Increased Heart Rate (Cardiac disorders) | 0 (0) | 1 (7)
Elevated Creatinine (Investigations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (10) | 2 (4)
Dizziness (Nervous system disorders) | 2 (3) | 1 (1)
Sinus Infection (Infections and infestations) | 1 (1) | 1 (1)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Slow Motor Function (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Drowsy (Nervous system disorders) | 2 (2) | 2 (3)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Head Burning Sensation (General disorders) | 0 (0) | 1 (1)
Ear Ache (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Jaw Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tooth Ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Head Cold (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Shaking (General disorders) | 0 (0) | 1 (1)
Left Arm Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left Scapula Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left Leg Fell Asleep (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right Arm Tingling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 1 (5) | 0 (0)
Temporal Bilateral Vein Throbbing (Nervous system disorders) | 1 (6) | 0 (0)
Increased Energy (General disorders) | 1 (1) | 0 (0)
Elevated ALT (Investigations) | 1 (1) | 0 (0)
Elevated AST (Investigations) | 1 (1) | 0 (0)
Thirsty (General disorders) | 2 (2) | 0 (0)
Excessive Sweating (General disorders) | 2 (4) | 0 (0)
Aching Leg Muscles (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Increased Urination (Renal and urinary disorders) | 1 (1) | 0 (0)
Sensations of Needles in Head (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cramping Sides (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Moody (Psychiatric disorders) | 1 (1) | 0 (0)
Calf Cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Light Sensitivity (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No